CLINICAL TRIAL: NCT00583492
Title: A Randomized, Controlled Trial of Replication-Competent Adenovirus-Mediated Suicide Gene Therapy in Combination With IMRT Versus IMRT Alone for the Treatment of Newly-Diagnosed Prostate Cancer With an Intermediate Risk Profile
Brief Title: Randomized Trial of Suicide Gene Therapy and Prostate Cancer
Acronym: ReCAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Benjamin Movsas, M.D., Chairman, Department of Radiation Oncology, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prostate4809
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Prostate Cancer
Keywords: Prostatic Neoplasms; Prostate Cancer; Adenocarinomas; Tumors of the Prostate; Gene Therapy; IMRT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ad5-yCD/mutTKSR39rep-ADP + IMRT (Experimental): Gene Therapy + IMRT
  Interventions: Biological: Ad5-yCD/mutTKSR39rep-ADP
- IMRT Alone (Active Comparator): IMRT: 40 x 2 Gy for a total dose of 80 Gy or 44 x 1.8 Gy for a total dose of 79.2 Gy
  Interventions: Radiation: IMRT

INTERVENTIONS:
Biological: Ad5-yCD/mutTKSR39rep-ADP — Ad5-yCD/mutTKSR39rep-ADP (1 x 10^12 vp) on day 1 Plus Radiation - 40 x 2 Gy for a total dose of 80 Gy or 44 x 1.8 Gy for a total dose of 79.2 Gy Plus 2 week course (weekdays only) of 5-FC and vGCV prodrug therapy
  Arms: Ad5-yCD/mutTKSR39rep-ADP + IMRT
Radiation: IMRT — 40 x 2 Gy for a total dose of 80 Gy or 44 x 1.8 Gy for a total dose of 79.2 Gy
  Arms: IMRT Alone

SUMMARY:
This is a randomized, controlled trial that will test the hypothesis that replication-competent adenovirus-mediated suicide gene therapy in combination with 80 Gy intensity modulated radiotherapy (IRMT)will improve freedom from failure (FFF) relative to 80 Gy IMRT alone in patients with newly-diagnosed prostate cancer with an intermediate-risk profile.

DETAILED DESCRIPTION:
OBJECTIVES

This is a randomized, controlled trial that will test the hypothesis that replication-competent adenovirus-mediated suicide gene therapy in combination with 80 Gy intensity modulated radiotherapy (IRMT)will improve freedom from failure (FFF) relative to 80 Gy IMRT alone in patients with newly-diagnosed prostate cancer with an intermediate-risk profile.

The trial contains two treatment arms:

Arm 1- Gene Therapy + IMRT Arm 2- IMRT

The study will be stratified by clinical site and pre-treatment risk factors (e.g., % positive biopsy cores, Gleason score.

* Gleason score 5/6 AND PSA <10 ng/mL; AND >=50% positive biopsy cores
* (Gleason score 5/6 and PSA 10-20 ng/mL) OR (Gleason score 7 and PSA 0 - 20 ng/mL); AND <50% positive biopsy cores
* Gleason score 5/6 and PSA 10-20 ng/mL) OR (Gleason score 7 and PSA 0-20 ng/mL) AND >=50% positive biopsy cores.

An interim safety analysis (Interim Analysis 1) will be conducted after the first 21 patients in the investigational therapy arm, and a total of 42 subjects in both arms, have completed the 90 day toxicity assessment following randomization (phase 2 component). If, at this point, there are no safety concerns as determined by the Data and Safety Monitoring Board (DSMB), the trial will continue as a phase 3 study with two additional interim analyses (Interim Analyses 2 & 3). The primary analysis for treatment efficacy will be based on all randomized subjects.

Primary

To assess the relative efficacy of replication-competent adenovirus-mediated suicide gene therapy in combination with 80 Gy intensity modulated radiotherapy (IMRT) versus 80 Gy IMRT alone in patients with newly-diagnosed prostate cancer with an intermediate-risk profile. The primary endpoint is freedom from failure (FFF) (biochemical or clinical).

Secondary

To assess the difference between the two treatment arms for:

* Acute (<= 90 days) and long-term (> 90 days) toxicity.
* Prostate biopsy status (12 cores) at 2 years.
* Freedom from distant metastases.
* Disease-specific and overall survival.
* Quality of life.

Exploratory

To examine:

* Possible effect of gene therapy on PSA doubling time (PSADT) after PSA failure.
* Possible association between the primary and secondary outcomes and Ad5-yCD/mutTKSR39rep-ADP adenovirus persistence (as measured by adenoviral DNA in blood).
* Possible association between the primary and secondary outcomes and specific immunological endpoints including levels of circulating CD4+ and CD8+ T lymphocytes, T-cell proliferation response, cytotoxic T lymphocyte (CTL) response, and development of antibodies to prostate-specific antigens.

ELIGIBILITY:
Inclusion Criteria:

* Men with histologically-confirmed adenocarcinoma of the prostate within 180 days prior to registration. To be eligible, the subjects must have one of the following conditions:

  * Stage T1 or T2, Gleason Score 7, PSA <= 20 ng/mL, Any number positive biopsy cores
  * Stage T1 or T2, Gleason Score 5 or 6, PSA >=10 ng/mL and <20 ng/mL, Any number positive biopsy cores
  * Stage T1 or T2, Gleason Score 5 or 6, PSA <10 ng/mL and >=50% positive biopsy cores
* Negative lymph nodes as established by imaging, nodal sampling, or dissection within 90 days prior to registration.
* No evidence of metastatic disease as evaluated by bone scan and CT scan of the abdomen and pelvis within 90 days prior to registration
* Karnofsky performance status >=70
* Subjects must have adequate baseline organ function, as assessed by the following laboratory values, within 30 days before initiating the study
* Adequate renal function with serum creatinine <=1.5 mg/dL or creatinine clearance >=45 mL/min/m2.
* Platelet count > 100,000/μL.
* Absolute neutrophil count > 1,000/μL.
* Hemoglobin > 10.0 g/dL.
* Normal partial thromboplastin time (PTT) and prothrombin (PT).
* Bilirubin < 1.5 mg/dL; SGOT and SGPT < 2.5 times upper limit of normal (ULN).
* Men of child-producing potential must be willing to consent to use effective contraception while on treatment and for at least 3 months afterwards.
* Subjects must possess the ability to give informed consent and express a willingness to meet all of the expected requirements of the protocol for the duration of the study.

Exclusion Criteria:

Subjects with the following conditions will be excluded from the study:

* Stage >= T3.
* Prostate specific antigen (PSA) > 20 ng/mL.
* Gleason score >= 8.
* Prostate volume >120cc.
* Pathologically positive lymph nodes or nodes > 1.5 cm on imaging. Note: nodes > 1.5 cm but biopsy negative are allowed.
* Evidence of M1 metastatic disease.
* Prior invasive malignancy except for non-melanoma skin cancer within 5 years of enrollment.
* Prognosis for survival of < 5 years.
* Prior radical prostatectomy, cryosurgery for prostate cancer, or bilateral orchiectomy for any reason.
* Prior radiotherapy, including brachytherapy, to the region of the study cancer that would result in overlap of radiation fields.
* Prior or planned androgen suppression therapy or prior systemic chemotherapy for the study cancer. Note that prior chemotherapy for a different cancer is allowed; however, patients must be >2 years post-completion of chemotherapy at time of registration. Patients on Proscar therapy must stop to be eligible.
* Severe, active co-morbidity defined as:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
* Transmural myocardial infarction within the last 6 months.
* Acute infection. Acute infection is defined by any viral, bacterial, or fungal infection that requires specific therapy within 72 hours of initiation of the study therapy.
* Positive serological test for HIV at baseline.
* Previous history of liver disease including hepatitis.
* Immunosuppressive therapy including systemic corticosteroids. Use of inhaled and topical corticosteroids is permitted.
* Impaired immunity or susceptibility to serious viral infections.
* Allergy to any product used in the protocol. (If the subject has an allergy to Ciprofloxacin, another antibiotic can be substituted at the discretion of the treating physician.
* Serious medical or psychiatric illness or concomitant medication, which, in the judgment of the principal investigator, might interfere with the subject's ability to respond to or tolerate the treatment or complete the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Movsas, M.D., Principal Investigator — Henry Ford Health System
Locations (2):
- United States (2):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan

REFERENCES:
- [Background] Freytag SO, Khil M, Stricker H, Peabody J, Menon M, DePeralta-Venturina M, Nafziger D, Pegg J, Paielli D, Brown S, Barton K, Lu M, Aguilar-Cordova E, Kim JH. Phase I study of replication-competent adenovirus-mediated double suicide gene therapy for the treatment of locally recurrent prostate cancer. Cancer Res. 2002 Sep 1;62(17):4968-76. PMID 12208748
- [Background] Freytag SO, Stricker H, Peabody J, Pegg J, Paielli D, Movsas B, Barton KN, Brown SL, Lu M, Kim JH. Five-year follow-up of trial of replication-competent adenovirus-mediated suicide gene therapy for treatment of prostate cancer. Mol Ther. 2007 Mar;15(3):636-42. doi: 10.1038/sj.mt.6300068. Epub 2007 Jan 16. PMID 17228316
- [Background] Freytag SO, Stricker H, Pegg J, Paielli D, Pradhan DG, Peabody J, DePeralta-Venturina M, Xia X, Brown S, Lu M, Kim JH. Phase I study of replication-competent adenovirus-mediated double-suicide gene therapy in combination with conventional-dose three-dimensional conformal radiation therapy for the treatment of newly diagnosed, intermediate- to high-risk prostate cancer. Cancer Res. 2003 Nov 1;63(21):7497-506. PMID 14612551
- [Background] Freytag SO, Movsas B, Aref I, Stricker H, Peabody J, Pegg J, Zhang Y, Barton KN, Brown SL, Lu M, Savera A, Kim JH. Phase I trial of replication-competent adenovirus-mediated suicide gene therapy combined with IMRT for prostate cancer. Mol Ther. 2007 May;15(5):1016-23. doi: 10.1038/mt.sj.6300120. Epub 2007 Mar 20. PMID 17375076
- [Result] Freytag SO, Stricker H, Lu M, Elshaikh M, Aref I, Pradhan D, Levin K, Kim JH, Peabody J, Siddiqui F, Barton K, Pegg J, Zhang Y, Cheng J, Oja-Tebbe N, Bourgeois R, Gupta N, Lane Z, Rodriguez R, DeWeese T, Movsas B. Prospective randomized phase 2 trial of intensity modulated radiation therapy with or without oncolytic adenovirus-mediated cytotoxic gene therapy in intermediate-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2014 Jun 1;89(2):268-76. doi: 10.1016/j.ijrobp.2014.02.034. Epub 2014 May 5. PMID 24837889

RESULTS

PARTICIPANT FLOW:
Groups:
- Gene Therapy + IMRT: Gene Therapy + IMRT
  Ad5-yCD/mutTKSR39rep-ADP: 1 x 10e12 sterile injectable solution, 1 injection on day one Plus Radiation - 40 x 2 Gy for a total dose of 80 Gy or 44 x 1.8 Gy for a total dose of 79.2 Gy Plus 2 week course (weekdays only) of 5-FC and vGCV prodrug therapy
Period: Overall Study
Arm/Group | Gene Therapy + IMRT | IMRT Alone
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gene Therapy + IMRT | IMRT Alone | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 13 | 14 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  United States | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Biochemical/Clinical Failure (FFF)
Description: Biochemical/Clinical Failure was defined as PSA nadir plus 2 ng/mL
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Gene Therapy + IMRT | IMRT Alone
Number analyzed (Participants) | 21 | 23
participants | 20 | 21

2. Secondary Outcome: Acute >= Grade 3 Treatment-related Toxicity
Description: This metric includes both expected and unexpected events Toxicities were graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 3
Time Frame: 90 days
Measure: Number; unit: percentage of adverse events
Arm/Group | Gene Therapy + IMRT | IMRT Alone
Number analyzed (Participants) | 21 | 23
percentage of adverse events | 4.6 | 6.0

3. Secondary Outcome: Positive Prostate Biopsy at 2 Years
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Gene Therapy + IMRT | IMRT Alone
Number analyzed (Participants) | 18 | 19
participants | 6 | 11

4. Secondary Outcome: Freedom From Distant Metastases
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Gene Therapy + IMRT | IMRT Alone
Number analyzed (Participants) | 21 | 23
participants | 21 | 23

5. Secondary Outcome: Disease-specific Survival
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Gene Therapy + IMRT | IMRT Alone
Number analyzed (Participants) | 21 | 23
participants | 21 | 23

6. Secondary Outcome: Decrease in Quality of Life
Description: Quality of Life was measured using the comprehensive Expanded Prostate Cancer Index Composite (EPIC) instrument 19 and 20
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Gene Therapy + IMRT | IMRT Alone
Number analyzed (Participants) | 21 | 23
participants | 0 | 0

ADVERSE EVENTS:
Groups:
- Gene Therapy + IMRT: Gene Therapy + IMRT
  Ad5-yCD/mutTKSR39rep-ADP: 1 x 10^12 sterile injectable solution, 1 injection on day one Plus Radiation - 40 x 2 Gy for a total dose of 80 Gy or 44 x 1.8 Gy for a total dose of 79.2 Gy Plus 2 week course (weekdays only) of 5-FC and vGCV prodrug therapy
Arm/Group | Gene Therapy + IMRT | IMRT Alone
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 21/21 | 7/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gene Therapy + IMRT (N=21) | IMRT Alone (N=23)
Flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 11 (11) | 2 (2) — Increased SGOT/SGPT
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 1 (1) — Low neutrophil counts
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 3 (3) — Low platelets

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No